CLINICAL TRIAL: NCT03525197
Title: Effects of a Whey Protein-based Multi-ingredient Supplement on Muscle Strength, Hypertrophy, and the Acute Satellite Cell Response, in Men and Women: a Double-blinded Randomized Controlled Trial
Brief Title: Effects of a Multi-ingredient Supplement Study: a Randomized Controlled Trial in Men and Women
Acronym: SRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HIREB 4449
Record Dates: First submitted 2018-04-27; First posted 2018-05-15 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Skeletal Muscle Hypertrophy
Keywords: Muscle Physiology; Nutrition

STUDY DESIGN:
Intervention Model Description: Parallel group design (with repeated measurements within each group)
Who Masked: Participant, Investigator
Masking Description: Each subject's supplement is coded with a different number, and neither the researchers nor the subjects are aware of the condition the subject is placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein-based supplement (Experimental): Participants in the experimental condition will consume a supplement containing Whey Protein Isolate (20g) and other ingredients
  Interventions: Dietary Supplement: Whey protein-based supplement
- Collagen protein-based supplement (Active Comparator): Participants in the experimental condition will consume a supplement containing Collagen protein (20g) and other ingredients
  Interventions: Dietary Supplement: Collagen protein-based supplement

INTERVENTIONS:
Dietary Supplement: Whey protein-based supplement — High quality protein supplement to be consumed twice daily
  Arms: Whey protein-based supplement
Dietary Supplement: Collagen protein-based supplement — Lower quality protein supplement to be consumed daily
  Arms: Collagen protein-based supplement

SUMMARY:
Resistance exercise training is a known stimulant for muscle protein synthesis (MPS) to occur, however the consumption of protein is also necessary to induce a shift towards a positive net protein balance. Other nutrients have been shown to be useful in the accretion of lean body mass and strength. Whey protein has been shown to improve muscle net protein balance after resistance exercise, more so when in conjunction with creatine. Furthermore, essential amino acids such as Leucine have been found to be important in moderating the shift towards a positive net protein balance, especially post-exercise and in combination with whey protein. Other vitamins and minerals have been shown to aid in permitting muscle protein synthesis rather than stimulating it, but are still necessary for optimal gains in hypertrophy. The effect of a multi-ingredient compound has rarely been investigated, and thus this study aims to combine whey protein, leucine, creatine, calcium citrate and vitamin D and test it in a resistance exercise training program over 12 weeks. Another novel aspect in this study will be testing this supplement against a placebo of equal amounts of protein and amino acids, the placebo will contain collagen protein and the non-essential amino acids alanine and glycine. Finally, this study will recruit both men and women (ages 18-30) to determine possible effects of the supplement on muscle hypertrophy in both sexes. We hypothesize that the synergistic effect of the ingredients in our supplement will induce hypertrophy to a larger degree than resistance exercise training with the placebo, and that these benefits will persist in both male and female participants.

DETAILED DESCRIPTION:
Supplementation in the form of whey protein, creatine and amino acids have all been shown to be a potent stimulus for muscle hypertrophy, when combined with resistance exercise. Burke et al. (2001) reported that males who supplemented with a combination of whey protein and creatine had greater increases in lean tissue mass and strength than those who supplemented with only whey protein or placebo. Hulmi at al. (2010) identified the most important component of whey to be its high concentration of the branched chain amino acid leucine, a critical amino acid for increasing muscle protein synthesis and suppressing muscle protein breakdown. The combination of leucine and whey protein has been shown to promote significant increases in muscle cross-sectional area. Vitamin D and calcium citrate have also been shown to enhance increases in muscle strength and lean mass, albeit in a permissive rather than stimulatory manner. Protein supplements have consistently been shown to promote greater gains in hypertrophy than their placebo counterparts, however these placebo supplements are often isoenergetic carbohydrate-based formulas. Few studies have compared two supplements with an equal amount of protein and amino acids, or have combined multiple beneficial ingredients to form a multicomponent supplement to promote greater gains in lean body mass and strength. Finally, sex differences in resistance training programs have rarely been studied, less so when testing a new supplement. Thus, the purpose of this study will be to determine whether there is an augmented effect of our nutritional supplement on the degree of hypertrophy in young male and female adults involved in a resistance training program. This nutritional supplement will be compared with a placebo containing an equivalent amount of collagen protein and non-essential amino acids. A secondary analysis will assess sex-based differences in strength and muscle size. Based on previous literature, we hypothesize that the combinatorial effect of whey protein, leucine, creatine, calcium citrate and vitamin D will induce hypertrophy to a larger degree than resistance exercise with the placebo in young adults.

A synergistic combination of ingredients with known benefits will be given twice daily to healthy young men and women (18-30 years old), (n = 22) in conjunction with a 12-week undulating periodized resistance training protocol, in which the repetition number and intensity of the training sessions will vary. Notable ingredients in this supplement include whey protein isolate (20g), leucine (2g), creatine monohydrate (2.5g), calcium citrate (300mg) and vitamin D (1000IU). The placebo condition, also comprised of males and females (18-30 years old), (n=22) will ingest a formulation containing an equivalent amount of collagen protein (20g), as well as an equivalent amount of amino acids (alanine, 1.4g and glycine, 0.6g). Pre- and post- assessments will include dual-energy x-ray absorptiometry (DEXA), one-rep maximum (1RM), and an ultrasound of the quadriceps. Four muscle biopsies will be taken from the vastus lateralis: 1) at rest prior to training, 2) 48h after an acute bout of exercise prior to training, 3) at rest post-training, and 4) 48h after an acute bout post-training. This allows for comparisons of acute and trained effects of both conditions. Using novel immunohistochemical staining procedures we will examine the resistance exercise-induced changes in fibre type distribution and fibre cross-sectional area in the supplement and placebo conditions as well as perform sex-based comparisons.

The novel aspect of this study will be the comparison of two isoenergetic, isonitrogenous supplements as stimulants for muscle protein accretion, as opposed to using carbohydrates as a placebo. The supplement will contain a new formulation of ingredients yet to be studied together. The synergistic effect of these ingredients will attempt to maximize muscle growth in both males and females, meaning that associations between sex and exercise can be assessed. This research will help us identify a new method to augment resistance exercise training through protein, amino acids, vitamins and minerals as well as expand the literature surrounding the effects of these ingredients on muscle hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years old
* Healthy based on questionnaire responses (see exclusion criteria)
* Recreationally active (exercising ~2x/week) with some resistance training experience (no more than 2 times weekly) allowed

Exclusion Criteria:

* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
* Arthritic conditions
* Individuals who consume any analgesic or anti-inflammatory drug(s), prescription or non-prescription, chronically will be excluded
* A history of neuromuscular complications
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Extensive history of resistance training in the year prior to study entry.
* Answers 'yes' to any question on the screening questionnaire

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Muscle Mass and fiber cross-sectional area | 10 weeks
  dual energy x-ray absorptiometry (DXA), ultrasound

SECONDARY OUTCOMES:
Satellite cell number, density, type I/type II fibre specific satellite cells and myonuclear domain | 10 weeks
  Histochemical methods will be used to determine how the supplement and training affect muscle growth and regenerative capacity, specifically the behaviour of satellite cells.
Strength | 10 weeks
  1RM testing pre- and post-training will be compared to determine how the supplement and training affect muscular strength
Fiber type distribution | 10 weeks
  Histochemical methods will be used to determine how the supplement and training affect fiber type distribution (% type I vs. % type II fibers pre- and post-training)

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Parise, PhD, Principal Investigator — McMaster University; Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario
  - Ivor Wynne Center, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] Burke DG, Chilibeck PD, Davidson KS, Candow DG, Farthing J, Smith-Palmer T. The effect of whey protein supplementation with and without creatine monohydrate combined with resistance training on lean tissue mass and muscle strength. Int J Sport Nutr Exerc Metab. 2001 Sep;11(3):349-64. doi: 10.1123/ijsnem.11.3.349. PMID 11591884
- [Background] Paddon-Jones D, Sheffield-Moore M, Zhang XJ, Volpi E, Wolf SE, Aarsland A, Ferrando AA, Wolfe RR. Amino acid ingestion improves muscle protein synthesis in the young and elderly. Am J Physiol Endocrinol Metab. 2004 Mar;286(3):E321-8. doi: 10.1152/ajpendo.00368.2003. Epub 2003 Oct 28. PMID 14583440
- [Background] Rondanelli M, Klersy C, Terracol G, Talluri J, Maugeri R, Guido D, Faliva MA, Solerte BS, Fioravanti M, Lukaski H, Perna S. Whey protein, amino acids, and vitamin D supplementation with physical activity increases fat-free mass and strength, functionality, and quality of life and decreases inflammation in sarcopenic elderly. Am J Clin Nutr. 2016 Mar;103(3):830-40. doi: 10.3945/ajcn.115.113357. Epub 2016 Feb 10. PMID 26864356
- [Background] Hulmi JJ, Lockwood CM, Stout JR. Effect of protein/essential amino acids and resistance training on skeletal muscle hypertrophy: A case for whey protein. Nutr Metab (Lond). 2010 Jun 17;7:51. doi: 10.1186/1743-7075-7-51. PMID 20565767
- [Background] Coburn JW, Housh DJ, Housh TJ, Malek MH, Beck TW, Cramer JT, Johnson GO, Donlin PE. Effects of leucine and whey protein supplementation during eight weeks of unilateral resistance training. J Strength Cond Res. 2006 May;20(2):284-91. doi: 10.1519/R-17925.1. PMID 16686554
- [Background] Tomlinson PB, Joseph C, Angioi M. Effects of vitamin D supplementation on upper and lower body muscle strength levels in healthy individuals. A systematic review with meta-analysis. J Sci Med Sport. 2015 Sep;18(5):575-80. doi: 10.1016/j.jsams.2014.07.022. Epub 2014 Aug 11. PMID 25156880
- [Background] Tang JE, Manolakos JJ, Kujbida GW, Lysecki PJ, Moore DR, Phillips SM. Minimal whey protein with carbohydrate stimulates muscle protein synthesis following resistance exercise in trained young men. Appl Physiol Nutr Metab. 2007 Dec;32(6):1132-8. doi: 10.1139/H07-076. PMID 18059587
- [Background] Verreijen AM, Verlaan S, Engberink MF, Swinkels S, de Vogel-van den Bosch J, Weijs PJ. A high whey protein-, leucine-, and vitamin D-enriched supplement preserves muscle mass during intentional weight loss in obese older adults: a double-blind randomized controlled trial. Am J Clin Nutr. 2015 Feb;101(2):279-86. doi: 10.3945/ajcn.114.090290. Epub 2014 Nov 26. PMID 25646324
- [Derived] Wageh M, Fortino SA, Pontello R, Maklad A, McGlory C, Kumbhare D, Phillips SM, Parise G. The Effect of Multi-Ingredient Protein versus Collagen Supplementation on Satellite Cell Properties in Males and Females. Med Sci Sports Exerc. 2024 Nov 1;56(11):2125-2134. doi: 10.1249/MSS.0000000000003505. PMID 39475860
- [Derived] Wageh M, Fortino SA, McGlory C, Kumbhare D, Phillips SM, Parise G. The Effect of a Multi-ingredient Supplement on Resistance Training-induced Adaptations. Med Sci Sports Exerc. 2021 Aug 1;53(8):1699-1707. doi: 10.1249/MSS.0000000000002641. PMID 33756525